CLINICAL TRIAL: NCT02033746
Title: A Crossover Study Using Transdermal Electroacupuncture as Adjunctive Treatment to Reduce Opiate Cravings in Post-Detox Outpatients Receiving Buprenorphine-Naloxone
Brief Title: Opiate Craving Reduction Study Using Post-detox Patients on Suboxone and Use of TEAS as Adjunctive Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Barbara MacIntyre MSN,RN, Barbara MacIntyre MSN,RN, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P001595
Record Dates: First submitted 2014-01-03; First posted 2014-01-13 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transdermal Electroacupuncture - Arm A (Experimental): week 1-2 real treatment, week 3-6 sham treatment with Han's Acupoint Nerve Stimulator while receiving concurrent buprenorphine-naloxone as prescribed
  Interventions: Device: Han's Acupoint Nerve Stimulator
- Transdermal Electroacupuncture - Arm B (Experimental): week 1-2 real treatment, week 3-6 sham treatment with Han's Acupoint Nerve Stimulator treatment while receiving concurrent buprenorphine-naloxone as prescribed
  Interventions: Device: Han's Acupoint Nerve Stimulator

INTERVENTIONS:
Device: Han's Acupoint Nerve Stimulator — frequency delivery(3 seconds of 2 Hz followed by 3 seconds of 100 Hz(dense disperse method).

SUMMARY:
Pilot study of 12 outpatients in early recovery from illicit drug use,post-detox and on buprenorphine-naloxone maintenance will be offered 12 TEAS adjunct treatments over 6 weeks(X2/week) to ascertain if they experience any improvement in mood,sleep,overall quality of life and decrease drug cravings ultimately while facing everyday life stressors.

DETAILED DESCRIPTION:
* this crossover study will involve participants who will be randomized into two treatment groups,A&B. TEAS treatments will be given for 30 minutes,X2/week,for 6 weeks(12total sessions). Group A will receive 2 weeks(4 sessions) of active treatment followed by 4 weeks of sham treatment(8 sessions). Group B will receive 2 weeks(4 sessions) of sham treatment,2 weeks (4 sessions)of real treatment,and finally 2 weeks (4 sessions) of sham treatment.
* parameters to be measured include vital signs and questionnaires weeks 1,3,5,6 to assess self-reported past 14-day substance use,alcohol and drug craving,withdrawal symptoms,sleep,mood,pain and overall quality of life.
* goals include better lives for post-detox opiate addicts as they incorporate this treatment into their lives,saving themselves and loved ones more horror,and their communities resources.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years old
* early recovery(0-3months of abstinence
* not currently detoxing
* maintained on buprenorphine-naloxone under the care of qualified MD
* proficient in the English language

Exclusion Criteria:

* having acute,psychiatric symptoms which would pose safety concerns,or an adherence to treatment barrier(active suicidality/psychosis/mania)
* severe cognitive disorders*not competent to give informed consent
* active cardiac disease or EKG abnormalities or with cardiac pacemaker
* currently detoxing from alcohol or illicit drugs
* inability or non-intention to attend all treatment sessions*history of seizures*pregnancy or breast feeding.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who attend all 12 Transdermal Electroacupuncture (TEAS) sessions | 6 weeks

SECONDARY OUTCOMES:
Number of participants who experience improvement in mood | 6 weeks
  Mood measured by self-report on the Quick Inventory of Depressive Symptomatology (QIDS-SR-16) questionnaire.
Number of participants who experience improvement in sleep | 6 weeks
  Sleep patterns measure by self report through the Pittsburgh Sleep Quality Index (PSQI) questionnaire
Number of participants who experience improvement in Quality-of-Life | 6 weeks
  Quality-of-Life measured by self-report through Short Form (SF)-36 questionnaire
Number of participants who report fewer cravings for drugs and alcohol | 6 weeks
  Cravings for drugs and alcohol measure by self-report through the Brief Addiction Monitor (BAM), the Craving Scale (CS), the Subjective Opiate Withdrawal Scale (SOWS), Substance Use Report, and a Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A MacIntyre, MSN,RN, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States